CLINICAL TRIAL: NCT05224921
Title: Study of Peripherel Perfusion Index to Predict Late Onset Sepsis in Very Low Birth Weight Infants
Brief Title: Peripherel Perfusion Index to Predict Sepsis in Very Low Birth Weight Infants
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-454
Record Dates: First submitted 2022-01-25; First posted 2022-02-04 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: VLBW - Very Low Birth Weight Infant
Keywords: Late onset sepsis; Peripheral perfusion index
MeSH Terms: interventions — Cohort Studies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Very low birth weight infants: Include very low birth weight infants admitted into NICU in Children's hospital of Fudan University, and prospectively observe whether they get late onset sepsis.
  Interventions: Other: Not applicable (cohort study)

INTERVENTIONS:
Other: Not applicable (cohort study) — This is a prospective observational study and does not include interventions. The exposure is peripheral perfusion index and the outcome is the incidence of late onset sepsis. From the day when the very low birth weight infant is admitted into hospital, PPI monitoring should be recorded once a day, and continuous monitoring would be recorded until 1 month after birth. Before collection, the infant will be confirmed to be in supine position with neutral temperature, and at the same time, the infant will be in a quiet state, without the contact and operation of medical personnel.

SUMMARY:
To explore the predictive value of peripheral perfusion index in late onset sepsis of very low birth weight infants , obtain the threshold by observing the perfusion index of very low birth-weight infants within one month after birth, this value can be used as a threshold to predict late onset sepsis in very low birth weight infants.

DETAILED DESCRIPTION:
From the day the very low birth weight infant was admitted to hospital, monitoring was recorded once a day, and continuous monitoring was recorded for 1 month. Before collection, the infant was confirmed to be in supine position with neutral temperature, and at the same time, the infant was in a quiet state, without the contact and operation of medical personnel. This study will first use LMS curve to fit the trend of perfusion index in very low birth weight infants within one month after birth.The perfusion index threshold of the outcome index was determined by ROC curve.

ELIGIBILITY:
Inclusion Criteria:

* Infants weighting <1500g
* Infants admitted to Children's Hospital of Fudan University

Ages: 0 Hours to 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infant's birth weight <1500g
Sampling Method: Probability Sample
Enrollment: 216 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of late onset sepsis | From admission into the ward to one month after birth
  Neonatal infection occurring 7 days after birth, confirmed by a doctor through laboratory positive indicators or clinical diagnosis

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No